CLINICAL TRIAL: NCT05200130
Title: The Effectiveness of Telerehabilitation With Self Mobilization in Patients With Subacromial Pain Syndrome
Brief Title: Effectiveness of Telerehabilitation on Subacromial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Erman Berk Celik, PT, Msc, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/074
Record Dates: First submitted 2021-12-07; First posted 2022-01-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Subacromial Pain Syndrome
Keywords: Pain; Functionality; Patient Satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home exercise group (Active Comparator): The home exercise program will be explained to the patients in the control group by the physiotherapist and the relevant brochures will be delivered to the patients. Home exercise program will take 30-45 min. İt will be applied 5 days a week for 8 weeks. Patients will receive a reminder message from the physiotherapist once a week.
  Interventions: Other: Home Exercise Group
- Manual Therapy Group (Active Comparator): Patients in the Manual Therapy Group will receive one-to-one physiotherapy sessions in the hospital 2 days a week for 8 weeks. In these sessions, soft tissue and joint mobilizations and exercises will be applied by physiotherapist.
  Interventions: Other: Manual Therapy Group
- Telerehabilitation Supported Group (Experimental): Telerehabilitation program will be applied 2 days a week for 8 weeks to patients in the telerehabilitation group. İt will take 30-45 min. A physiotherapist will meet with patients via videoconferencing over the internet and guide the program.
  Interventions: Other: Telerehabilitation Group

INTERVENTIONS:
Other: Home Exercise Group — The home exercise program includes an educational training program and posture correction exercises. The program includes stretching and strengthening exercises of the neck and shoulder complex.
  Arms: Home exercise group
Other: Manual Therapy Group — Manual Therapy includes deep friction massage and myofascial relaxation techniques to shoulder and neck complex, active and resistant shoulder complex movements, shoulder complex mobilization, mobilization cervical joints.
  The home exercise program includes an educational training program and posture correction exercises. The program includes stretching and strengthening exercises of the neck and shoulder complex.
  Arms: Manual Therapy Group
Other: Telerehabilitation Group — The telerehabilitation program applied to the same home exercise group. In addition, to the home exercises, these patients will apply active mobilization called self-mobilization. Self-myofascial release, active glenohumeral joint mobilization, thoracic mobilization, and active cervical mobilization.
  Arms: Telerehabilitation Supported Group

SUMMARY:
The aim of this study is to evaluate the effectiveness of supervised exercise therapy with active soft tissue and joint mobilization.

The effectiveness of telerehabilitation- active mobilization and exercises in the evaluation of pain and function in patients with subacromial pain syndrome will be examined and compared with face-to-face treatment, which is passive manual therapy.

DETAILED DESCRIPTION:
Shoulder pain is common in the population. Various treatment modalities are used. Due to the Coronavirus disease (COVID-19), the problems in patients' access to hospitals and rehabilitation services caused telerehabilitation to be on the agenda. Telerehabilitation can be summarized as the delivery of rehabilitation services to those in need by using communication technologies. This method covers the steps of evaluation, monitoring, prevention, intervention, control, training, and consultation. In addition, as a new treatment application, its effectiveness will be measured in patients with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-50 who complain of shoulder pain
* Individuals diagnosed with a partial tear of the rotator cuff smaller than 1 cm and As a result of the examination performed by the physician stage 1 or 2 subacromial impingement syndrome.
* Two of the following tests are positive Hawkins-Kennedy, painful arc or infraspinatus muscle strength tests
* Presence of shoulder pain lasting longer than 6 weeks that limits activity.
* Being literate and not having cognitive dysfunction.

Exclusion Criteria:

* Presence of other orthopedic, neurological and systemic problems affecting the neck, shoulder and back complex,
* Patients with heart failure and using a pacemaker,
* Labral tears and other intraarticular structural pathologies
* Signs of adhesive capsulitis
* Grade 3 or full thickness rotator cuff tear
* BMİ > 30 kg/m
* Having been included in a physical therapy program related to the same side shoulder joint in the last 1 year
* Using non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 8 weeks and 12 weeks | Change from Baseline in Pain at 8 weeks and 12 weeks
  Visual Analog Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain.
Change from Baseline in Short-Form Mcgill Pain questionnaire (SF-MPQ) at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  The McGill Pain questionnaire will be used to evaluate a person experiencing significant pain..
  The pain rating index has 2 subscales:
  1. Sensory subscale with 11 words
  2. Affective subscale with 4 words from the original MPQ. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe.
Change from Baseline in Posture Analysis at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  Corbin posture analysis will be used. This form include lateral and posterior analyzes. Physiotherapist marks between 0 = none 3= severe point to disorders. Total score will calculate excellent = 0-2 to Poor = 12 or more
Change from Baseline in range of motion of the shoulder at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  Range of motion of the shoulder will be evaluated with a standard goniometer.
Kibler classification for changes in position and scapular movements at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  Kibler classification will be use assessment of Scapular Dyskinesia. Identifying changes in position and scapular movements that predispose to shoulder injuries. Identifying the type of abnormal scapular movement: type I, type II and type III.
Lateral Scapular Slide test at 8 weeks and 12 weeks | Change from Baseline in Lateral Scapulara Slide at 8 weeks and 12 weeks
  Lateral Scapular Slide test will be use assessment of Scapular Dyskinesia. The Measurement should not vary more than 1 to 1.5 cm, more the 1.5 cm difference significant.
Change from Baseline in Glenohumeral internal rotation deficit (GIRD) at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  GIRD is a condition resulting in the loss of internal rotation of the glenohumeral joint as compared to the contralateral side.
Change from Baseline in Disabilities of the Arm, Shoulder, and Hand (QuickDASH) at 8 weeks and 12 weeks | Baseline, 8 weeks, and 12 weeks
  QuickDASH will be used for assessing functional ability of the patients. The QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
Change from Baseline in The Shoulder Pain and Disability Index (SPADI)at 8 weeks and 12 weeks | Baseline, 8 weeks, 12 weeks
  The SPADI will be used to assess shoulder pain and dysfunction. It consists of 13 items that assess two different areas. The first five items measure the pain, and the next eight items assess patient's disability.
Patient Satisfaction questionnaire at 8 weeks. | 8 weeks
  The Patient Satisfaction questionnaire will be used to assess the patient's satisfaction with the treatment received. Patient Satisfaction questionnaire (PSQ) contains 18 items tapping each of the seven dimensions of satisfaction with medical care measured by the PSQ-18.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation
Locations (1):
- Erman Berk Celik, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celik EB, Tuncer A. Comparing the Efficacy of Manual Therapy and Exercise to Synchronized Telerehabilitation with Self-Manual Therapy and Exercise in Treating Subacromial Pain Syndrome: A Randomized Controlled Trial. Healthcare (Basel). 2024 May 24;12(11):1074. doi: 10.3390/healthcare12111074. PMID 38891149